CLINICAL TRIAL: NCT04985058
Title: Real-world Clinical Outcome and Toxicity Data in Patients With Breast Cancer Treated With Abemaciclib Combined With Endocrine Therapy: the Experience of the Hellenic Cooperative Oncology Group
Brief Title: Real-world Data in Patients With Breast Cancer Treated With Abemaciclib
Acronym: ENDURANCE
Status: Recruiting | Type: Observational
Sponsor: Hellenic Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: RWD_abemaciclib
Record Dates: First submitted 2021-07-26; First posted 2021-08-02 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer
Keywords: abemaciclib; real-world data
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with breast cancer randomised in arm A of digital platform: Patients with breast cancer treated with abemaciclib in combination with endocrine treatment and randomised in Arm A of the digital platform. Patients randomised in arm A will receive a an acknowledgement and suggestion to stay in contact with their clinician.
- Patients with breast cancer randomised in arm B of digital platform: Patients with breast cancer treated with abemaciclib in combination with endocrine treatment and randomised in Arm B of the digital platform. Patients randomised in arm A will receive a an acknowledgement and suggestion to stay in contact with their clinician; additionally they will receive personalised support (as a few word text) for each side-effect reported.

SUMMARY:
The present study will assess real-world clinical outcomes and adverse events from treatment with endocrine therapy combined with abemaciclib in patients with HR-positive, HER2-negative advanced breast cancer.

DETAILED DESCRIPTION:
Protocol was amended in November 2021, after the recent FDA approval of abemaciclib in the adjuvant setting. On October 12, 2021, FDA approved abemaciclib with endocrine therapy for the adjuvant treatment of adult patients with hormone receptor -positive, HER2-negative, node-positive, early breast cancer at high risk of recurrence and a Ki-67 score ≥20%. Our study will now include real-world data on efficacy and toxicity of abemaciclib in the adjuvant setting as well. 2-negative advanced breast cancer. Patients who are enrolled and the patients to be enrolled will refer to a dedicated online platform (CARE ACROSS platform) where they can register their side-effects of cancer and the treatment received at frequent intervals. Patients will be randomized in the platform in two arms with an allocation 1:1(automatically by the platform). After every report of their side-effects, patients in Arm A will receive an acknowledgement and suggestion to stay in contact with their clinician. After every report of their side- effects, patients in Arm B will receive an acknowledgment and suggestion to stay in contact with their clinician; additionally they will receive personalised support (as a few word text) for each side-effect reported. Clinicians involved in the trial will refer patients (upon enrollment or to those already enrolled) to a dedicated online platform. Patients will sign up by entering their patient ID and their email address (and picking their password for security).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed HR-positive, HER2-negative breast cancer
* Treated at Hellenic Cooperative Oncology Group (HeCOG)-affiliated departments of oncology
* 18 years or older
* Any menopausal status
* Treatment with abemaciclib in combination with endocrine therapy
* Any endocrine therapy
* At least two months of treatment with abemaciclib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically confirmed HR-positive, HER2-negative breast cancer treated with abemaciclib in combination with endocrine therapy
Sampling Method: Non-Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2021-10-06 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Through the completion of the study, for an average of 6 months
  the time from treatment initiation to either the first documented disease progression or death from any cause

SECONDARY OUTCOMES:
Overall survival | From date of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 96 months
  The time from treatment initiation to patient death or last contact
Efficacy of the digital support through personalised support in patients with BC | Up to 30 months
Toxicity rate | Up to 30 months
  Adverse events from the time from treatment initiation to disease progression, patient death or last contact

CONTACTS AND LOCATIONS:
Locations (1):
- Hellenic Oncology Cooperative Group, Athens, Greece

REFERENCES:
- [Derived] Fountzilas E, Aravantinou-Fatorou E, Dadouli K, Economopoulou P, Tryfonopoulos D, Vernadou A, Vorrias E, Vagionas A, Nikolaidi A, Karageorgopoulou S, Koumarianou A, Boukovinas I, Mauri D, Kokkali S, Christopoulou A, Tsoukalas N, Assi A, Spathas N, Kosmidis P, Koutras A, Fountzilas G, Psyrri A. Real-World Toxicity and Effectiveness Study of Abemaciclib in Greek Patients with Hormone Receptor-Positive/Human Epidermal Growth Factor Receptor 2-Negative Breast Cancer: A Multi-Institutional Study. Cancers (Basel). 2025 Jul 31;17(15):2543. doi: 10.3390/cancers17152543. PMID 40805239